CLINICAL TRIAL: NCT03400189
Title: Preliminary Pilot Exploration of the Pharmacokinetic and Tolerability Profile of Sulthiame in Healthy Volunteers
Brief Title: Pharmacokinetics and Tolerability of Sulthiame
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire Vaudois (Other)
Collaborators: Advicenne Pharma (Industry)
Responsible Party: Principal Investigator, Thierry Buclin, Professor, Centre Hospitalier Universitaire Vaudois
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: C01CS
Record Dates: First submitted 2017-12-14; First posted 2018-01-17 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy | interventions — sulthiame

STUDY DESIGN:
Intervention Model Description: Phase I, single centre, prospective, ascending single oral doses, open-label, 3-period clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): Single oral dose of sulthiame (Ospolot® tablets)
  * Period I: 50 mg
  * Period II: 100 mg
  * Period III: 200 mg given 3 weeks apart
  Interventions: Drug: Sulthiame

INTERVENTIONS:
Drug: Sulthiame — Single dose (50, 100, 200 mg)
  Other Names: Ospolot

SUMMARY:
This preliminary pilot exploration aims at specifying the pharmacokinetic parameters of sulthiame, formulated as an immediate release tablet, thus helping to design proper clinical trials for the future assessment of new paediatric formulations currently under development. The clinical tolerability to single doses of sulthiame will also be closely monitored to orient future trials.

DETAILED DESCRIPTION:
Sulthiame (or sultiame), marketed in the 60's in Germany, Austria, Switzerland, Israel, Australia and Japan under the brand name Ospolot®, has progressively become the therapeutic first choice in benign focal epilepsies of childhood in these countries.

Its antiepileptic activity is thought to result from the inhibition of various subtypes of carbonic anhydrase (hCA), in particular cytosolic hCA II, thus inducing a degree of intracellular acidification sufficient to stabilize seizure-eliciting neurons. The pharmacokinetic profile of sulthiame was scarcely studied in humans.

Sulthiame is a suitable candidate for paediatric formulation optimization, as the current formulation (coated tablets of 50 or 200 mg) allows neither precise and adapted dosing, nor convenient administration to young children.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male subjects aged between 18 and 45 years.
2. Body weight (BW) ranging between 55 and 95 kg, providing body mass index (BMI) is between 18 and 29 kg/m2
3. Absence of significant findings in the medical history and physical examination as judged by the Investigator, especially for cardiovascular, pulmonary, haematological and nervous systems
4. Absence of significant laboratory abnormalities as judged by the Investigator. Gilbert's syndrome (increased total and unconjugated bilirubin when fasting) will be accepted if mild
5. Absence of clinically significant abnormalities on 12-lead electrocardiogram (ECG)
6. Negative urine drug screen (amphetamines, benzodiazepines, cannabis, cocaine, opiates)
7. Commitment to refrain from travels outside Europe over the whole study duration.
8. Ability to understand the procedures, agreement to participate and willingness to give written informed consent
9. Co-operative attitude and availability for scheduled visits over the entire study period.

Exclusion Criteria:

1. History of major cardiovascular, pulmonary, hepatic, immunological, renal, haematological, gastrointestinal, genitourinary, neurological, or rheumatologic disorders
2. Active diseases of any type, including inflammatory disorders and infections. Mild acne is permissible providing no systemic or local treatment is provided or planned (except for cleaning lotions)
3. History of significant allergy or asthma. Allergic rhinitis or conjunctivitis is acceptable if non symptomatic when starting the study and if symptoms are not anticipated to occur during the study to a point that would require corticosteroid therapy (e.g. in case of annual use)
4. History of cardiovascular dysfunction if considered as clinically relevant (conduction abnormality, arrhythmia, bradycardia, angina pectoris, cardiac hypertrophy unless elicited by training, pulmonary embolism)
5. Hypertension defined as supine blood pressure >150/90 mmHg or recurrent hypotensive events considered as clinically relevant or documented orthostatic hypotension
6. Sick sinus syndrome, known long QT syndrome, reproducible observation of QTc >440 msec or of pronounced sinus bradycardia (<40 bpm/min)
7. Intense sport activities. Moderate sport is acceptable and activities should remain fairly constant throughout the study
8. Any clinically significant laboratory value on screening that are not within normal range on single repeat (Gilbert's syndrome acceptable if mild)
9. Positive hepatitis B & C antigen screen
10. Positive HIV antibody screen or screen not performed
11. Any recent acute illness or sequelae thereof which could expose the subject to a higher risk or might confound the results of the study
12. Treatment in the previous three months with any drug known to have well-defined potential for toxicity to a major organ
13. History of hypersensitivity to any drug if considered as serious including sulthiame or the excipients of the study formulation
14. Use of any medication the week prior to study or as based on 5 plasma half-life rule and throughout study, including aspirin or other over-the-counter (OTC) preparation. Paracetamol is permissible before and during study as a concomitant medication but only with Investigator's permission.
15. Participation in a clinical investigation or blood donation of 500 ml within the past 3 months
16. History of relevant alcohol or drug abuse
17. Smoking. Consumption of <5 cigarettes/day or equivalent is acceptable providing the subject can refrain from smoking from one week before and during the whole study duration
18. Consumption of a large quantity of coffee, tea, chocolate (more than 4 cups/day) or equivalent (Cola drinks)
19. Present consumption of a large quantity of alcohol or wine (>0.5 L wine/day) or equivalent, (equivalent to more than >48 g ethanol per day).
20. Project to conceive a child during the study period (by principle of precaution, while no indication exists for a definite reproductive risk following paternal exposure)
21. Psychological status which could impact on subject's ability to give informed consent
22. Any feature of subject's medical history or present condition which, in the Investigator's opinion, could confound the results of the study, complicate its interpretation, or represent a potential risk for the subject.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2018-02-12 (Actual); Primary Completion 2018-05-22 (Actual); Study Completion 2018-08-30 (Actual)

PRIMARY OUTCOMES:
Elimination half-life of sultiame after single doses of 50, 100 and 200 mg of sulthiame in 4 healthy volunteers. | 9 weeks
  Sultiame plasma concentration will be measured at predefined times after dose administration, the results will be plotted graphically and traditional pharmacokinetic calculations (log-linear regression) will be used to derive estimates of this pharmacokinetic parameter. This is a descriptive outcome and no statistical test is applied.
Area Under curve (AUC) of sultiame after single doses of 50, 100 and 200 mg of sulthiame in 4 healthy volunteers. | 9 weeks
  Sultiame plasma concentration will be measured at predefined times after dose administration, the results will be plotted graphically and traditional pharmacokinetic calculations (numerical integration through trapezoidal rule) will be used to derive estimates of this pharmacokinetic parameter. This is a descriptive outcome and no statistical test is applied.
Systemic drug clearance of sultiame after single doses of 50, 100 and 200 mg of sulthiame in 4 healthy volunteers. | 9 weeks
  Sultiame concentration will be measured at predefined times after dose administration, the results will be plotted graphically and traditional pharmacokinetic calculations (ratio of administered dose over AUC) will be used to derive estimates of this pharmacokinetic parameter. This is a descriptive outcome and no statistical test is applied.
Distribution volume of sultiame after single doses of 50, 100 and 200 mg of sulthiame in 4 healthy volunteers. | 9 weeks
  Sultiame plasma concentration will be measured at predefined times after dose administration, the results will be plotted graphically and traditional pharmacokinetic calculations (product of clearance by half-life divided by the logarithm of 2) will be used to derive estimates of this pharmacokinetic parameter. This is a descriptive outcome and no statistical test is applied.

SECONDARY OUTCOMES:
Dose linearity of plasma exposure to sultiame | 9 weeks
  A linear regression model will be applied to AUC as a function of dose, and the conclusion of dose linearity will be accepted if the model appears statistically non-inferior to an ANOVA model.
Plasma free fraction of sultiame | 9 weeks
  The ratios of free over total plasma concentrations, and of whole blood over total plasma concentrations will be calculated, and its stability over the range of concentrations will be checked by statistical analysis for trend.
Erythrocyte binding of sultiame | 9 weeks
  The ratios of free over total plasma concentrations, and of whole blood over total plasma concentrations will be calculated, and its stability over the range of concentrations will be checked by statistical analysis for trend.
Validation of a liquid chromatography-mass spectrometry (LC-MS/MS) assay method for the determination of sultiame in biological fluids | 9 weeks
  The analytical method used for the study will be assessed for its sensitivity (estimation of detection and quantification limits), precision (estimation of intra-day and inter-day reproducibility) and accuracy (estimation of sultiame recovery using spiked samples). The analytical method will be considered validated if all criteria are within the acceptance range set by FDA/ICH recommendations.

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Clinical Pharmacology, Lausanne, Canton of Vaud, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided